CLINICAL TRIAL: NCT01555944
Title: Screening and Management of Cardiovascular Risk in Belgian Women Aged > or = 65 Years With Metastatic Breast Cancer Before and After Anthracycline Treatment
Brief Title: Prospective Observational Study in Patients With Metastatic Breast Cancer Treated With Anthracyclines
Status: Completed | Type: Observational
Sponsor: Teva Pharma (Industry)
Responsible Party: Sponsor
Other Study IDs: MyCard
Record Dates: First submitted 2012-03-14; First posted 2012-03-16 (Estimated); Last update posted 2016-04-25 (Estimated); Status verified 2016-04

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is an open, multicentre, prospective observational (non-interventional) study, performed in Belgium.

Principal objectives:

1. To evaluate the prevalence of cardiovascular risk factors and cardiac function (as routinely evaluated) before treatment with anthracyclines of patients with metastatic breast cancer (MBC) aged > or = 65 years
2. To observe the management of cardiovascular risk during and after anthracycline treatment
3. To compare liposomal versus non-liposomal anthracycline therapy (ratio 1:1) on cardiac function, outcome and quality of life (EORTC QLQ-C30)

Secondary objectives:

1. To evaluate the efficacy of anthracyclines on progression free survival and tumor response as routinely measured (e.g. recist criteria, tumor markers and other exams)
2. To evaluate cardiovascular event type: ECG changes, arrhythmia, decrease of ejection fraction, heart failure and rate according to allocated treatment.
3. To find out how quality of life, e.g. such as described according to EORTC QLQ-C30 criteria or Karnofsky index is achieved in the various patient subgroups
4. To correlate the therapeutic choice and posology of anthracyclines for MBC with Cardiovascular risk at baseline
5. To calculate the cardiovascular risk according to SCORE

DETAILED DESCRIPTION:
The physician will be requested:

* To include 15 consecutive patients aged > or = 65 years who will be treated with anthracyclines in first and second line MBC. The physician will be encouraged to enrol 2 arms of 8 patients (one treated with liposomal and one with non-liposomal anthracyclines) for observation and comparison. Each arm will be closed as soon as 150 patients are included at a national level.
* To report their cardiovascular risk factors
* To provide the results of routinely performed cardiac evaluation before treatment
* To monitor routinely cardiovascular parameters during treatment and report them afterwards
* To monitor efficacy and tolerance of treatments, as normal practice prescribes, reported and related to the variables described in objectives
* To ensure that quality of life will be assessed with the EORTC QLQ-C30 questionnaire
* To monitor and report progression free survival and cardiac events
* To record and transmit spontaneously reported adverse events. These will be handled according to legal requirements

Follow-up will cover a period of 15 months following inclusion.

The study will have 3 visits and 2 contacts:

* One visit at entry
* One visit after 3 cycles of anthracycline containing therapy
* One visit at the end of treatment
* Contact at 9 months after inclusion
* Contact at 15 months after inclusion

It is planned to include data from 15 consecutive female patients per specialized center in Belgium.

The total number of patients aimed is 300.

ELIGIBILITY:
Inclusion Criteria:

* women aged 65 years old or more
* with confirmed metastatic breast cancer (MBC)
* who will be treated with anthracyclines in first or second line
* who have a Karnofsky score at baseline of 50
* who agree and are able to fill in the EORTC QLQ-C30 questionnaire
* who gave their informed consent

Exclusion Criteria:

* women having contra-Indications for anthracyclines
* women aged < 65 years old
* with no metastatic breast cancer
* who will not be eligible for an anthracycline treatment in first or second line MBC
* who have a Karnofsky less than 50
* who disagree or are unable to fill in the EORTC QLQ-C30 questionnaire
* women refusing or not having signed their informed consent

Min Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Belgian women aged > or = 65 years with metastatic breast cancer before and after anthracycline treatment.
  Patients will be included in 24 centers specialized in the treatment of breast cancer, in Belgium.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2012-02; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
cardiovascular risk factors | 15 months

CONTACTS AND LOCATIONS:
Overall Officials: Christel Fontaine, MD, Principal Investigator — Universitair Ziekenhuis Brussel
Locations (24):
- Belgium (24):
  - ZNA Middelheim, Antwerp
  - Cliniques du Sud Lux - St Joseph, Arlon
  - Imelda, Bonheiden
  - Clinique Saint-Luc, Bouge
  - AZ KLINA, Brasschaat
  - AZ St Jan, Bruges
  - CHU Brugmann, Brussels
  - Erasme, Brussels
  - UZ Brussel, Brussels
  - CHIREC - Centre Hospitalier Interrégional Edith Cavell, Brussels
  - CSF, Chimay
  - AZ St-Maarten, Duffel
  - UZA, Edegem
  - AZ St-Dimpna, Geel
  - AZ St-Lucas, Ghent
  - ZNA Jan Palfijn, Merksem
  - CHR, Namur
  - CMSE, Namur
  - AZ Damiaan, Ostend
  - Clinique St Pierre, Ottignies
  - AZ Nikolaas, St-Niklaas
  - Centre Hospitalier de Wallonie picarde - site IMC, Tournai
  - CHPLT, Verviers
  - CHU Mont-Godinne, Yvoir

IPD SHARING:
Plan to Share IPD: No